CLINICAL TRIAL: NCT01392300
Title: Prospective, Double-blind, Placebo-controlled, Randomized, Multi-center Study With an Open-label Extension Period to Investigate the Efficacy and Safety of NT 201 in the Treatment of Post-stroke Spasticity of the Upper Limb
Brief Title: Efficacy and Safety Study of Botulinum Toxin Type A Against Placebo to Treat Spasticity in the Arm After a Stroke
Acronym: PURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRZ 60201/SP/3001; 2010-023043-15 (EudraCT Number)
Record Dates: First submitted 2011-07-07; First posted 2011-07-12 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2016-11

CONDITIONS: Post-stroke Spasticity of the Upper Limb
MeSH Terms: interventions — incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DB IncobotulinumtoxinA (Xeomin) (400 U) (Experimental): IncobotulinumtoxinA (Xeomin) (400 Units): Main period, one injection session - double-blind (DB), randomized treatment assignment
  Interventions: Drug: IncobotulinumtoxinA (400 Units)
- DB Placebo Comparator (Placebo Comparator): Placebo to incobotulinumtoxinA (Xeomin) (400 Units): Main period, one injection session - double-blind (DB), randomized treatment assignment
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: IncobotulinumtoxinA (400 Units) — Main period: One injection session of solution, prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl), 400 units, total volume 8.0 mL; Mode of administration: intramuscular injection
  Other Names: Xeomin
  Arms: DB IncobotulinumtoxinA (Xeomin) (400 U)
Drug: Placebo Comparator — Main period: one injection session of solution, prepared by reconstitution of powder with 0.9% NaCl, corresponding total placebo volume 8.0 mL; Mode of administration: intramuscular injection
  Arms: DB Placebo Comparator

SUMMARY:
The purpose of this study is to determine whether injections of Botulinum toxin type A into muscles of the upper limb are effective in treating spasticity in patients after stroke.

DETAILED DESCRIPTION:
The study consists of a randomized, double-blind, placebo-controlled, parallel-group, single-dose main period followed by an open-label, non-controlled, repeated-dose extension period (Open-Label Extension Period - OLEX).

ELIGIBILITY:
Inclusion Criteria:

* Upper limb spasticity
* Time since stroke greater than 3 months
* Need for 400 U Botulinum toxin type A

Exclusion Criteria:

* Body weight below 50kg
* Fixed contractures of the upper limb
* Generalized disorders of muscle activity like Myasthenia gravis that preclude use of Botulinum toxin Type A
* Infection at the injection site

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2011-09; Primary Completion 2013-03 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — Merz Pharmaceuticals GmbH
Locations (47):
- United States (13):
  - Merz Investigational Site #001184, Downey, California
  - Merz Investigational Site #001017, Fountain Valley, California
  - Merz Investigational Site #001188, Miami, Florida
  - Merz Investigational Site #001037, Augusta, Georgia
  - Merz Investigational Site #001186, Chicago, Illinois
  - Merz Investigational Site # 001110, Overland Park, Kansas
  - Merz Investigational Site #001198, Stratford, New Jersey
  - Merz Investigational Site #001240, Chapel Hill, North Carolina
  - Merz Investigational Site #001009, Winston-Salem, North Carolina
  - Merz Investigational Site #001241, Philadelphia, Pennsylvania
  - Merz Investigational Site #001211, Pittsburgh, Pennsylvania
  - Merz Investigational Site #001245, Chattanooga, Tennessee
  - Merz Investigational Site #001226, Houston, Texas
- Czechia (8):
  - Merz Investigational Site #420046, Brno
  - Merz Investigational Site #420029, Brno
  - Merz Investigational Site #420028, Olomouc
  - Merz Investigational Site #420024, Ostrava-Poruba
  - Merz Investigational Site #420025, Pardubice
  - Merz Investigational Site #420030, Prague
  - Merz Investigational Site #420045, Prague
  - Merz Investigational Site #420047, Rychnov nad Kněžnou
- Merz Investigational Site #049134, Rostock, Germany
- Hungary (4):
  - Merz Investigational Site #036004, Budapest
  - Merz Investigational Site # 036009, Budapest
  - Merz Investigational Site #036005, Nyíregyháza
  - Merz Investigational Site #036008, Szeged
- India (7):
  - Merz Investigational Site #091003, Porur, Chennai
  - Merz Investigational Site #091006, Bangalore, Karnataka
  - Merz Investigational Site #091002, Trivandrum, Kerala
  - Merz Investigational Site #091004, New Delhi, New Delhi
  - Merz Investigational Site #091007, Chennai, Tamil Nadu
  - Merz Investigational Site #091008, Coimbatore, Tamil Nadu
  - Merz Investigational Site #091001, Lucknow, Uttar Pradesh
- Poland (10):
  - Merz Investigational Site # 048029, Gdansk
  - Merz Investigational Site #048044, Kielce
  - Merz Investigational Site #048031, Krakow
  - Merz Investigational Site #048050, Lodz
  - Merz Investigational Site #048051, Lublin
  - Merz Investigational Site #048032, Olsztyn
  - Merz Investigational Site #048053, Poznan
  - Merz Investigational Site #048023, Warsaw
  - Merz Investigational Site #048052, Warsaw
  - Merz Investigational Site #048033, Warsaw
- Russia (4):
  - Merz Investigational Site #007010, Krasnoyarsk
  - Merz Investigational Site #007011, Moscow
  - Merz Investigational Site #007009, Saint Petersburg
  - Merz Investigational Site #007005, Stavropol

REFERENCES:
- [Result] Elovic EP, Munin MC, Kanovsky P, Hanschmann A, Hiersemenzel R, Marciniak C. Randomized, placebo-controlled trial of incobotulinumtoxina for upper-limb post-stroke spasticity. Muscle Nerve. 2016 Mar;53(3):415-21. doi: 10.1002/mus.24776. Epub 2015 Dec 15. PMID 26201835
- [Derived] Marciniak C, Munin MC, Brashear A, Rubin BS, Patel AT, Slawek J, Hanschmann A, Hiersemenzel R, Elovic EP. IncobotulinumtoxinA Treatment in Upper-Limb Poststroke Spasticity in the Open-Label Extension Period of PURE: Efficacy in Passive Function, Caregiver Burden, and Quality of Life. PM R. 2020 May;12(5):491-499. doi: 10.1002/pmrj.12265. Epub 2020 Jan 22. PMID 31647185
- [Derived] Marciniak C, Munin MC, Brashear A, Rubin BS, Patel AT, Slawek J, Hanschmann A, Hiersemenzel R, Elovic EP. IncobotulinumtoxinA Efficacy and Safety in Adults with Upper-Limb Spasticity Following Stroke: Results from the Open-Label Extension Period of a Phase 3 Study. Adv Ther. 2019 Jan;36(1):187-199. doi: 10.1007/s12325-018-0833-7. Epub 2018 Nov 27. PMID 30484117

RESULTS

PARTICIPANT FLOW:
Groups:
- Double-blind IncobotulinumtoxinA (Xeomin) (400 Units): IncobotulinumtoxinA (Xeomin) (400 Units): Main period, one injection session - double-blind, randomized treatment assignment
- Double-blind Placebo Comparator: Placebo to incobotulinumtoxinA (Xeomin) (400 Units): Main period, one injection session - double-blind, randomized treatment assignment
- OLEX IncobotulinumtoxinA (Xeomin) (400 Units, 3 Injections): IncobotulinumtoxinA (Xeomin) (400 Units): OLEX period, three injection sessions - open-label treatment assignment
Period: Main Period (MP)
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator | OLEX IncobotulinumtoxinA (Xeomin) (400 Units, 3 Injections)
Started | 210 | 107 | 0
Completed | 199 | 100 | 0
Not Completed | 11 | 7 | 0
Not completed — Predefined discontinuation criteria | 2 | 3 | 0
Not completed — Withdrawal by Subject | 5 | 1 | 0
Not completed — Lost to Follow-up | 3 | 3 | 0
Not completed — Non-compliance | 1 | 0 | 0
Period: Open Label Extension (OLEX) Period
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator | OLEX IncobotulinumtoxinA (Xeomin) (400 Units, 3 Injections)
Started | 0 (Subjects from double-blind arms were switched to arm OLEX IncobotulinumtoxinA (Xeomin) (...)) | 0 (Subjects from double-blind arms were switched to arm OLEX IncobotulinumtoxinA (Xeomin) (...)) | 299 (Subjects from double-blind arms were switched to arm OLEX IncobotulinumtoxinA (Xeomin) (...))
Completed | 0 | 0 | 248
Not Completed | 0 | 0 | 51
Not completed — Protocol Violation | 0 | 0 | 13
Not completed — Lack of Efficacy | 0 | 0 | 3
Not completed — Non-compliance | 0 | 0 | 1
Not completed — Death | 0 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 17
Not completed — Lost to Follow-up | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Population: Safety evaluation set (The subset of all subjects who were exposed to investigational product in the main period)
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator | Total
Number analyzed (Participants) | 210 | 107 | 317
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (11.9) | 57.8 (10.9) | 56.1 (11.6)
Gender [Count of Participants; unit: Participants]
  Female | 120 | 61 | 181
  Male | 90 | 46 | 136
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 22 | 12 | 34
  Unknown or Not Reported | 184 | 95 | 279
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 27 | 13 | 40
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 3 | 9
  White | 175 | 91 | 266
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 26 | 12 | 38
  Czech Republic | 46 | 25 | 71
  Hungary | 23 | 9 | 32
  Poland | 66 | 38 | 104
  Russian Federation | 22 | 10 | 32
  Germany | 1 | 0 | 1
  India | 26 | 13 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Ashworth Scale (AS) Score of Primary Target Clinical Pattern
Description: Primary target clinical pattern was defined by investigator for each subject at baseline visit and was either flexed wrist or clenched fist or flexed elbow.
  The Ashworth Scale is well known and commonly used in clinical trials with spasticity. It was used to categorize severity of spasticity by judging resistance to passive movement. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension).
Time Frame: Week 4
Population: Full Analysis set (all subjects who were randomized after the Amended Protocol Version 3.0, dated 11-MAY-2012 became effective, who were treated, and for whom at least an AS baseline value for the primary target clinical pattern is given). Missing values were imputed by the last observation carried forward (LOCF) approach.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.9 (0.06) | -0.5 (0.08)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.7 to -0.3], Standard Error of Mean 0.1

2. Primary Outcome: Investigator's Global Impression of Change
Description: This is the co-primary outcome measure. The Global Impression of Change Scale [GICS] is used to measure the investigator's impression of change due to treatment. The response option is a common 7-point Likert scale that ranges from -3 = very much worse to +3 = very much improved.
Time Frame: Week 4
Population: Full Analysis set (all subjects who were randomized after the Amended Protocol Version 3.0, dated 11-MAY-2012 became effective, who were treated, and for whom at least an AS baseline value for the primary target clinical pattern is given). Missing values were imputed by zero change (worst case).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | 1.2 (0.07) | 0.9 (0.09)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.003, ANCOVA; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [0.1 to 0.5], Standard Error of Mean 0.11

3. Secondary Outcome: Response Rates on the Ashworth Scale at Week 4 Calculated for the Primary Target Clinical Pattern
Description: Primary target clinical pattern was defined by investigator for each subject at baseline visit and was either flexed wrist or clenched fist or flexed elbow. Subjects with a reduction of one point were defined as responder for the aim of the efficacy analysis.
Time Frame: Week 4
Population: Full Analysis set (all subjects who were randomized after the Amended Protocol Version 3.0, dated 11-MAY-2012 became effective, who were treated, and for whom at least an AS baseline value for the primary target clinical pattern is given). Missing values were imputed by worst case (=non-responder).
Measure: Number; unit: participants
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
participants | 119 | 33
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.28, 95% CI 2-sided [2.43 to 7.52]

4. Secondary Outcome: Response Rates on the Ashworth Scale at Week 8 Calculated for the Primary Target Clinical Pattern
Description: as for outcome 3
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
participants | 104 | 34
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.69, 95% CI 2-sided [1.56 to 4.63]

5. Secondary Outcome: Response Rates on the Ashworth Scale at Week 12 Calculated for the Primary Target Clinical Pattern
Description: as for outcome 3
Time Frame: Week 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
participants | 68 | 22
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.004, Regression, Logistic; Odds Ratio (OR) = 2.48, 95% CI 2-sided [1.33 to 4.61]

6. Secondary Outcome: Response Rates on the Ashworth Scale at Week 4 Calculated for the Muscle Group Flexed Wrist
Description: The Ashworth Scale is well known and commonly used in clinical trials with spasticity. It was used to categorize severity of spasticity by judging resistance to passive movement. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension). Subjects with a reduction of one point were defined as responder for the aim of the efficacy analysis.
Time Frame: Week 4
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
participants | 102 | 31
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.13, 95% CI 2-sided [1.76 to 5.57]

7. Secondary Outcome: Response Rates on the Ashworth Scale at Week 8 Calculated for the Muscle Group Flexed Wrist
Description: as for outcome 6
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
participants | 90 | 33
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.021, Regression, Logistic; Odds Ratio (OR) = 1.92, 95% CI 2-sided [1.10 to 3.34]

8. Secondary Outcome: Response Rates on the Ashworth Scale at Week 12 Calculated for the Muscle Group Flexed Wrist
Description: as for outcome 6
Time Frame: Week 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
participants | 59 | 17
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 2.58, 95% CI 2-sided [1.32 to 5.05]

9. Secondary Outcome: Response Rates on the Ashworth Scale at Week 4 Calculated for the Muscle Group Flexed Elbow
Description: as for outcome 6
Time Frame: Week 4
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
participants | 99 | 28
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.72, 95% CI 2-sided [2.06 to 6.72]

10. Secondary Outcome: Response Rates on the Ashworth Scale at Week 8 Calculated for the Muscle Group Flexed Elbow
Description: as for outcome 6
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
participants | 85 | 28
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 2.50, 95% CI 2-sided [1.40 to 4.46]

11. Secondary Outcome: Response Rates on the Ashworth Scale at Week 12 Calculated for the Muscle Group Flexed Elbow
Description: as for outcome 6
Time Frame: Week 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
participants | 52 | 21
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.102, Regression, Logistic; Odds Ratio (OR) = 1.70, 95% CI 2-sided [0.90 to 3.22]

12. Secondary Outcome: Response Rates on the Ashworth Scale at Week 4 Calculated for the Muscle Group Clenched Fist
Description: as for outcome 6
Time Frame: Week 4
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
participants | 90 | 26
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.95, 95% CI 2-sided [1.67 to 5.23]

13. Secondary Outcome: Response Rates on the Ashworth Scale at Week 8 Calculated for the Muscle Group Clenched Fist
Description: as for outcome 6
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
participants | 82 | 27
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 2.46, 95% CI 2-sided [1.37 to 4.41]

14. Secondary Outcome: Response Rates on the Ashworth Scale at Week 12 Calculated for the Muscle Group Clenched Fist
Description: as for outcome 6
Time Frame: Week 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
participants | 49 | 19
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.069, Regression, Logistic; Odds Ratio (OR) = 1.87, 95% CI 2-sided [0.95 to 3.69]

15. Secondary Outcome: Response Rates on the Ashworth Scale at Week 4 Calculated for the Muscle Group Thumb-in-palm
Description: as for outcome 6
Time Frame: Week 4
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
participants | 56 | 21
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.034, Regression, Logistic; Odds Ratio (OR) = 2.05, 95% CI 2-sided [1.05 to 4.00]

16. Secondary Outcome: Response Rates on the Ashworth Scale at Week 8 Calculated for the Muscle Group Thumb-in-palm
Description: as for outcome 6
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
participants | 52 | 23
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.169, Regression, Logistic; Odds Ratio (OR) = 1.61, 95% CI 2-sided [0.82 to 3.16]

17. Secondary Outcome: Response Rates on the Ashworth Scale at Week 12 Calculated for the Muscle Group Thumb-in-palm
Description: as for outcome 6
Time Frame: Week 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
participants | 35 | 20
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.920, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.49 to 2.18]

18. Secondary Outcome: Response Rates on the Ashworth Scale at Week 4 Calculated for the Muscle Group Pronated Forearm
Description: as for outcome 6
Time Frame: Week 4
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
participants | 73 | 19
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.56, 95% CI 2-sided [1.83 to 6.91]

19. Secondary Outcome: Response Rates on the Ashworth Scale at Week 8 Calculated for the Muscle Group Pronated Forearm
Description: as for outcome 6
Time Frame: Week 8
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
participants | 64 | 20
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.007, Regression, Logistic; Odds Ratio (OR) = 2.41, 95% CI 2-sided [1.28 to 4.56]

20. Secondary Outcome: Response Rates on the Ashworth Scale at Week 12 Calculated for the Muscle Group Pronated Forearm
Description: as for outcome 6
Time Frame: Week 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
participants | 51 | 15
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.018, Regression, Logistic; Odds Ratio (OR) = 2.26, 95% CI 2-sided [1.15 to 4.41]

21. Secondary Outcome: Changes From Baseline to Week 4 in Ashworth Scale Score for Treated Muscle Group Flexed Wrist.
Description: The Ashworth Scale is well known and commonly used in clinical trials with spasticity. It was used to categorize severity of spasticity by judging resistance to passive movement. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension).
Time Frame: Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.8 (0.06) | -0.5 (0.08)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.5 to -0.2]

22. Secondary Outcome: Changes From Baseline to Week 8 in Ashworth Scale Score for Treated Muscle Group Flexed Wrist.
Description: as for outcome 21
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.6 (0.06) | -0.4 (0.08)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.011, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to -0.1], Standard Error of Mean 0.09

23. Secondary Outcome: Changes From Baseline to Week 12 in Ashworth Scale Score for Treated Muscle Group Flexed Wrist.
Description: as for outcome 21
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.3 (0.05) | -0.1 (0.07)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.032, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.3 to 0.0], Standard Error of Mean 0.08

24. Secondary Outcome: Changes From Baseline to Week 4 in Ashworth Scale Score for Treated Muscle Group Flexed Elbow.
Description: as for outcome 21
Time Frame: Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.7 (0.05) | -0.3 (0.07)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.6 to -0.2], Standard Error of Mean 0.08

25. Secondary Outcome: Changes From Baseline to Week 8 in Ashworth Scale Score for Treated Muscle Group Flexed Elbow.
Description: as for outcome 21
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.6 (0.05) | -0.3 (0.07)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.5 to -0.1], Standard Error of Mean 0.09

26. Secondary Outcome: Changes From Baseline to Week 12 in Ashworth Scale Score for Treated Muscle Group Flexed Elbow.
Description: as for outcome 21
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.4 (0.05) | -0.2 (0.07)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.029, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.3 to 0.0], Standard Error of Mean 0.08

27. Secondary Outcome: Changes From Baseline to Week 4 in Ashworth Scale Score for Treated Muscle Group Clenched Fist.
Description: as for outcome 21
Time Frame: Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.7 (0.06) | -0.3 (0.08)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.5 to -0.2], Standard Error of Mean 0.09

28. Secondary Outcome: Changes From Baseline to Week 8 in Ashworth Scale Score for Treated Muscle Group Clenched Fist.
Description: as for outcome 21
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.6 (0.05) | -0.4 (0.08)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.019, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to 0.0], Standard Error of Mean 0.09

29. Secondary Outcome: Changes From Baseline to Week 12 in Ashworth Scale Score for Treated Muscle Group Clenched Fist.
Description: as for outcome 21
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.3 (0.05) | -0.1 (0.07)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.137, ANCOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.3 to 0.0], Standard Error of Mean 0.08

30. Secondary Outcome: Changes From Baseline to Week 4 in Ashworth Scale Score for Treated Muscle Group Thumb-in-palm.
Description: as for outcome 21
Time Frame: Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.4 (0.05) | -0.2 (0.07)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.013, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to 0.0], Standard Error of Mean 0.09

31. Secondary Outcome: Changes From Baseline to Week 8 in Ashworth Scale Score for Treated Muscle Group Thumb-in-palm.
Description: as for outcome 21
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.3 (0.05) | -0.2 (0.08)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.131, ANCOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.3 to 0.0], Standard Error of Mean 0.09

32. Secondary Outcome: Changes From Baseline to Week 12 in Ashworth Scale Score for Treated Muscle Group Thumb-in-palm.
Description: as for outcome 21
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.2 (0.05) | -0.1 (0.07)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.714, ANCOVA; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.08

33. Secondary Outcome: Changes From Baseline to Week 4 in Ashworth Scale Score for Treated Muscle Group Pronated Forearm.
Description: as for outcome 21
Time Frame: Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.5 (0.05) | -0.2 (0.07)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.5 to -0.2], Standard Error of Mean 0.08

34. Secondary Outcome: Changes From Baseline to Week 8 in Ashworth Scale Score for Treated Muscle Group Pronated Forearm.
Description: as for outcome 21
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.4 (0.05) | -0.2 (0.07)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.008, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to -0.1], Standard Error of Mean 0.09

35. Secondary Outcome: Changes From Baseline to Week 12 in Ashworth Scale Score for Treated Muscle Group Pronated Forearm.
Description: as for outcome 21
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.3 (0.05) | -0.1 (0.07)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.062, ANCOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.3 to 0.0], Standard Error of Mean 0.08

36. Secondary Outcome: Changes From Baseline to Week 4 in Disability Assessment Scale - Principal Therapeutic Target Domain
Description: The Disability Assessment Scale consists of the four domains hygiene, dressing, limb position, and pain which were assessed on a 4-point scale with the values 0 (=no disability), 1 (=mild disability), 2 (=moderate disability), and 3 (=severe disability).
Time Frame: Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.5 (0.05) | -0.3 (0.07)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.006, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to -0.1], Standard Error of Mean 0.08

37. Secondary Outcome: Changes From Baseline to Week 8 in Disability Assessment Scale - Principal Therapeutic Target Domain
Description: as for outcome 36
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.5 (0.05) | -0.3 (0.07)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.076, ANCOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.3 to 0.0], Standard Error of Mean 0.08

38. Secondary Outcome: Changes From Baseline to Week 12 in Disability Assessment Scale - Principal Therapeutic Target Domain
Description: as for outcome 36
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.4 (0.05) | -0.4 (0.06)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.416, ANCOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.08

39. Secondary Outcome: Changes From Baseline to Week 4 in Disability Assessment Scale - Domain Hygiene
Description: as for outcome 36
Time Frame: Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.4 (0.05) | -0.1 (0.06)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.4 to -0.1], Standard Error of Mean 0.07

40. Secondary Outcome: Changes From Baseline to Week 8 in Disability Assessment Scale - Domain Hygiene
Description: as for outcome 36
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.4 (0.05) | -0.2 (0.07)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.175, ANCOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.3 to 0.1], Standard Error of Mean 0.08

41. Secondary Outcome: Changes From Baseline to Week 12 in Disability Assessment Scale - Domain Hygiene
Description: as for outcome 36
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.3 (0.05) | -0.1 (0.07)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.140, ANCOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.3 to 0.0], Standard Error of Mean 0.08

42. Secondary Outcome: Changes From Baseline to Week 4 in Disability Assessment Scale - Domain Dressing
Description: as for outcome 36
Time Frame: Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.4 (0.05) | -0.2 (0.06)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.007, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to -0.1], Standard Error of Mean 0.07

43. Secondary Outcome: Changes From Baseline to Week 8 in Disability Assessment Scale - Domain Dressing
Description: as for outcome 36
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.4 (0.05) | -0.2 (0.07)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.018, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.3 to 0.0], Standard Error of Mean 0.08

44. Secondary Outcome: Changes From Baseline to Week 12 in Disability Assessment Scale - Domain Dressing
Description: as for outcome 36
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.3 (0.04) | -0.1 (0.06)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.105, ANCOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.3 to 0.0], Standard Error of Mean 0.07

45. Secondary Outcome: Changes From Baseline to Week 4 in Disability Assessment Scale - Domain Limb Position
Description: as for outcome 36
Time Frame: Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.5 (0.05) | -0.3 (0.07)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.016, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to 0.0], Standard Error of Mean 0.08

46. Secondary Outcome: Changes From Baseline to Week 8 in Disability Assessment Scale - Domain Limb Position
Description: as for outcome 36
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.4 (0.05) | -0.2 (0.07)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.014, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.4 to 0.0], Standard Error of Mean 0.08

47. Secondary Outcome: Changes From Baseline to Week 12 in Disability Assessment Scale - Domain Limb Position
Description: as for outcome 36
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.4 (0.05) | -0.3 (0.06)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.220, ANCOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.07

48. Secondary Outcome: Changes From Baseline to Week 4 in Disability Assessment Scale - Domain Pain
Description: as for outcome 36
Time Frame: Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.2 (0.06) | -0.2 (0.08)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.429, ANCOVA; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to 0.1], Standard Error of Mean 0.09

49. Secondary Outcome: Changes From Baseline to Week 8 in Disability Assessment Scale - Domain Pain
Description: as for outcome 36
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.2 (0.06) | -0.2 (0.08)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.884, ANCOVA; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.09

50. Secondary Outcome: Changes From Baseline to Week 12 in Disability Assessment Scale - Domain Pain
Description: as for outcome 36
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator
Number analyzed (Participants) | 171 | 88
units on a scale | -0.3 (0.06) | -0.2 (0.09)
Statistical Analysis 1: Comparison: Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) vs Double-blind Placebo Comparator; Test type: Superiority or Other; p = 0.844, ANCOVA; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.10

ADVERSE EVENTS:
Time Frame: From the timepoint of first injection until 12 weeks +/- 3 days after last injection
Description: The investigator asked the patient for AEs systematically at each visit.
Groups:
- OLEX IncoboutulinumtoxinA (Xeomin) (400 Units, 3 Injections): IncobotulinumtoxinA (Xeomin) (400 Units): OLEX period, three injection sessions - open-label treatment assignment
Arm/Group | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) | Double-blind Placebo Comparator | OLEX IncoboutulinumtoxinA (Xeomin) (400 Units, 3 Injections)
Serious Adverse Events (participants affected / at risk) | 7/210 | 2/107 | 22/296
Other Adverse Events (participants affected / at risk) | 6/210 | 4/107 | 32/296
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) (N=210) | Double-blind Placebo Comparator (N=107) | OLEX IncoboutulinumtoxinA (Xeomin) (400 Units, 3 Injections) (N=296)
Pneumonia (Infections and infestations) | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0
Peipheral ischaemia (Vascular disorders) | 2 | 0 | 0
Pancreatic enlargement (Gastrointestinal disorders) | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 2
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cardiac death (General disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Pseudobulbar palsy (Nervous system disorders) | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind IncobotulinumtoxinA (Xeomin) (400 Units) (N=210) | Double-blind Placebo Comparator (N=107) | OLEX IncoboutulinumtoxinA (Xeomin) (400 Units, 3 Injections) (N=296)
Headache (Nervous system disorders) | 1 (1) | 3 (6) | 3 (6)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 8 (9)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 8 (10)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 7 (9)
Epilepsy (Nervous system disorders) | 5 (6) | 0 (0) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.